CLINICAL TRIAL: NCT03033433
Title: An Open-label Phase I Study to Assess the Safety and Tolerability Profile of Three Escalating Doses of DCB-DM101 in Healthy Volunteers and Optimum Dose of DCB-DM101 as add-on Treatment in Type 2 Diabetes Mellitus (T2DM) Patients
Brief Title: DCB-DM101 in Healthy Volunteers and for Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VitNovo, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCB-DM101-CP001
Record Dates: First submitted 2016-12-25; First posted 2017-01-26 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2016-12

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Masking Description: open label
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DCB-DM101, 500 mg tablet, determination of optimal dose (Experimental): Stage 1:Dose level 1(1 tablet of DCB-DM101 q.d. for 7 days orally);Dose level 2(2 tablets of DCB-DM101 q.d. for 7 days orally);Dose level 3(4 tablets of DCB-DM101 q.d. for 7 days orally) Stage 2:Optimum dose of DCB-DM101 determined in Stage 1 as add-on treatment in T2DM patients for 14 days, q.d., orally
  Interventions: Drug: DCB-DM101

INTERVENTIONS:
Drug: DCB-DM101 — determination of optimal dose for Stage 2

SUMMARY:
An Open-Label Phase I Study to Assess the Safety and Tolerability Profile of Three Escalating Doses of DCB-DM101 in Healthy Volunteers and Optimum Dose of DCB-DM101 as Add-on Treatment in Type 2 Diabetes Mellitus (T2DM) Patients

DETAILED DESCRIPTION:
This is a single center, open-label, phase-I study consisting of two stages: Stage 1 will be dose-escalation study to assess the safety and tolerability profile of three escalating doses of DCB-DM101 in healthy volunteers and Stage 2 will apply optimum dose of DCB-DM101 as add-on treatment in T2DM patients. In Stage 2, patients are allowed to receive metformin for T2DM for routine use of which the dosing regimen should not be adjusted. No other medication/treatments for T2DM are allowed. Stage 2 can only be proceeded upon the approval of health authority in Taiwan. After determining the optimal dose for Stage 2, the reasons for determining such dose together with relevant supporting data should be submitted to health authority in Taiwan for review and to determine whether stage 2 can be proceeded and which dose should be employed for stage 2.

ELIGIBILITY:
Inclusion Criteria:

Stage 1

1. Adult, male or female aged between 20-40 years old;
2. Physically and mentally healthy subjects as confirmed by an interview, medical history, clinical examination, chest X-rays, and electrocardiogram;
3. Body Mass Index (BMI) between 18.5 and 24, inclusive, (BMI will be calculated as weight in kilogram [kg]/height in meters2 [m2]);
4. Clinically normal hematology, biochemistry and urinalysis determinations based on investigator's discretion;
5. Subject is willing and able to comply with study procedures and sign informed consent.

Stage 2

1. Male or female aged between 20-70 years old;
2. Diagnosed T2DM (WHO 1999 criteria);
3. Not effective in alleviating T2DM after monotherapy of metformin 1,500mg/day [or 1,000mg/day if unable to tolerate higher dose] for 3 months
4. HbA1c of 7.0 % to 9.0% (inclusive);
5. BMI of at most 35 kg/m2;
6. Subject is willing and able to comply with study procedures and sign informed consent

Exclusion Criteria:

Stage 1

1. Subjects who have a history or evidence of a medical condition that would expose them to an undue risk of a significant adverse event or interfere with the assessments of safety or pharmacodynamics variables during the course of the trial, including but not limited to hepatic, renal, respiratory, cardiovascular, endocrine, immune, neurological, musculoskeletal or hematological disease as determined by the clinical judgment of the investigator;
2. Subject has received any investigational agent within 28 days or 5 half-lives, whichever is longer, prior to the first dose of study drug;
3. Subjects have taken or potentially take any prescription medication and/or over the-counter medication from within 1 week prior to the first dose of study drug to the end of study period;
4. Subject has alcohol, caffeine, grapefruit juice, or nicotine consumption within 24 hours prior to the administration of study drug;
5. Female subject of childbearing potential who: is lactating; or has positive urine pregnancy test at Visit 1; or refuses to adopt at least two forms of birth control (at least one of which must be a barrier method) during the study.

Stage 2

1. Known or suspected allergy to any ingredients of study product
2. Pregnant or lactating or premenopausal with childbearing potential but not taking at least two forms of birth control (at least one of which must be a barrier method) during the study.

Note: Acceptable forms include:

1. Established use of oral, injected or implanted hormonal methods of contraception.
2. Placement of an intrauterine device (IUD) or intrauterine system (IUS).
3. Barrier methods of contraception: Condom OR Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository. 3. Participated in another clinical trial and received an investigational drug within four weeks prior to the present trial
4. Impaired hepatic function defined as alanine aminotransferase (ALT), aspartate transaminase (AST) or alkaline phosphatase (ALP) at least 2.5 times upper referenced limit
5. Impaired renal function defined as serum-creatinine at least 1.3 mg/dL (at least 115 umol/L) for males and at least 1.2 mg/dL (at least 106 umol/L) for females
6. With any uncontrolled illness or a history of any illness judged by the investigator that entering the trial may be detrimental to the subject
7. Metformin contraindications according to the package insert
8. Current treatment with systemic corticosteroids.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Stage 1: Optimal dose for Stage 2, dose limiting toxicity (DLT) | 7 months
  Primary endpoint, DLT is defined as: Any causally related adverse event as judged by investigator is greater than or equal to Grade 2. The causality of each adverse event to investigational product will be judged by investigator during the conduction of each dosing cohort in Stage I. DSMB will reevaluate the causality of each DLT after the completion or termination of this dosing cohort judged by investigator to determine whether dose escalation or entering to stage 2 can be proceeded.Optimal Dose will be one tablet or two tablets or 4 tablets. the optimal dose for stage 2 is defined using rules as follows but will be determined by sponsor and investigators.
Stage 2: Number of Participants with Adverse events and Serious adverse events that are related to treatment | 3 months
  Specified:Primary endpoint, An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a study medication and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a study medication, whether or not related to the study medication.
  A Serious Adverse Event is defined as an AE meeting one of the following conditions. Death during the period of protocol defined surveillance. Life threatening Event defined as a participant at immediate risk of death at the time of the event. An event requiring inpatient hospitalization or prolongation of existing hospitalization during the period of protocol defined surveillance. Results in congenital anomaly or birth defect. Results in a persistent or significant disability and incapacity.

SECONDARY OUTCOMES:
Stage1: Number of Participants with Adverse events and Serious adverse events that are related to treatment | 7 months
  Secondary endpoint, An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a study medication and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a study medication, whether or not related to the study medication.
  A Serious Adverse Event is defined as an AE meeting one of the following conditions. Death during the period of protocol defined surveillance. Life threatening Event defined as a participant at immediate risk of death at the time of the event. An event requiring inpatient hospitalization or prolongation of existing hospitalization during the period of protocol defined surveillance. Results in congenital anomaly or birth defect. Results in a persistent or significant disability and incapacity.
Stage2: Change from baseline in results of oral glucose tolerance test (OGTT) | 0 (pre-dose) and 0.5, 1, 1.5, 2, 2.5 hours post-dose
  While patient takes OGTT at Screening visit, blood glucose will be monitor at right before, 0.5, 1, 1.5, and 2 hr after administration of solution containing 75 g glucose. While at visit 2 and 4, blood glucose will be monitored at pre-dose, right before taking solution containing 75 g glucose(30 mins after dosing), 1, 1.5, 2, and 2.5 hr after administration of dose.
Stage2: Change from baseline in biomarker( serum insulin) testing results. | Visits 1 (-30 to 1 days), Visit 2 (Day 1), Visits 3 (Day 8), Visit 4(Day 14)and 5 (Day 28).
  Biomarker consists of serum insulin. Insulin will be measured at all the same time points where blood glucose is measured including OGTT test time points for Visits 1 (-30 to 1 days), 2 (Day 1), and 4(Day 14), and single blood sampling besides laboratory test for Visits 3 (Day 8) and 5 (Day 28).
Stage2: Change from baseline in biomarker( serum fructosamine) testing results. | Visit 1 (-30 to 1 days), Visit 3 (Day 8), Visit 4 (Day 14), and Visit 5 (Day 28).
  Fructosamine at will be measured at Visit 1 (-30 to 1 days), Visit 3 (Day 8), Visit 4 (Day 14), and Visit 5 (Day 28).

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Jen Hung, MD, Principal Investigator — Tri-Service General Hospital
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No